CLINICAL TRIAL: NCT06298864
Title: Digital Cognitive Behavioral Therapy for Cardiac Anxiety Following Acute Coronary Syndrome: a Randomized Controlled Trial Comparing CBT to a Digital Lifestyle Intervention
Brief Title: Internet-based Behavioral Intervention Following ACS
Acronym: ACS-CBT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Josefin Särnholm, PhD, Lic. Psychologist, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASC-RCT 2
Record Dates: First submitted 2024-02-26; First posted 2024-03-07 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Acute Coronary Syndrome; Online CBT Targeting Cardiac Anxiety
Keywords: Cardiac Anxiety; Acute Coronary Syndrome; ACS; Internet-CBT; CBT; Secondary prevention
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based Cognitive Behavioral Therapy (Internet-CBT) (Experimental): Internet-CBT following ACS is exposure-based, centering on exposure to cardiac related symptoms and situations. The CBT is therapist-guided and lasts for 8 weeks.
  Interventions: Behavioral: Internet-CBT
- Internet-based Cardiac Lifestyle intervention (Internet-CL) (Active Comparator): Internet-CL is based on strategies for behavioral change and guidelines on health promoting lifestyle modifications following ACS. The Internet-CL is therapist-guided and lasts for 8 weeks.
  Interventions: Behavioral: Internet-CL

INTERVENTIONS:
Behavioral: Internet-CBT — * Common reactions following ACS. The role of cardiac anxiety and avoidance behavior on quality of life and physical health. Brief training in self-observation, i.e., labeling. General lifestyle advice on e.g., physical activity, diet.
  * Identifying life areas impaired by ACS-related disability or symptom fear. Set health behavioral goals i.e., increased physical activity and gradually take steps towards them.
  * Gradual exposure to physical sensations (e.g., palpitations due to physical activity) to reduce fear of these symptoms.
  * Gradual exposure to avoided situations, activities and increase in physical activity.
  * Prevention of relapse into avoidance behaviors by identifying risk situations and conduct a plan forward on maintaining a healthy physically and active lifestyle.
  Arms: Internet-based Cognitive Behavioral Therapy (Internet-CBT)
Behavioral: Internet-CL — * Education on ACS, risk factors, its treatments and medication.
  * Education and advice promoting healthy habits regarding diet, alcohol and tobacco.
  * Education and advice regarding physical activity and the beneficial effects on health.
  * Education regarding common emotional reactions following ACS.
  * Prevention of relapse and plan forward to maintain a healthy lifestyle.
  Arms: Internet-based Cardiac Lifestyle intervention (Internet-CL)

SUMMARY:
The aim of this study is to evaluate if an online Cognitive Behavioral Therapy (CBT) protocol customized for patients following Acute Coronary Syndrome (ACS), reduce cardiac anxiety, enhance Quality of Life (QoL), and promote increased physical activity while controlling for caregiver attention, utilizing an active control group receiving internet-based cardiac lifestyle intervention.

DETAILED DESCRIPTION:
ACS is a leading global cause of mortality and health-related losses. Following ACS, many individuals exhibit symptoms of anxiety and depression, recognized risk factors for recurrent cardiovascular events. Specifically, anxiety related to cardiac symptoms and avoidance behavior, known as cardiac anxiety, has been shown to increase the long-term risk of adverse cardiac events.

The purpose of the present interdisciplinary research project is to develop and evaluate an online CBT protocol tailored for ACS patients. This project comprises a series of clinical studies aimed at accumulating knowledge about the most effective ways to treat ACS patients with CBT over the internet.

The aim of this study is to assess whether internet-based CBT, following ACS, reduces cardiac anxiety and improves QoL, while controlling for caregiver attention and expectancy of improvement using an active control group.

Method: A randomized controlled trial is conducted where participants are randomly assigned to either internet-based CBT (N= 88) or internet-based cardiac lifestyle intervention (internet-CL) (N= 88). The active control group receives internet-CL, focusing on lifestyle modification and health-promoting behaviors. Weekly therapist support through online written communication is provided to participants in both groups. Both treatment are conducted over 8-weeks and are comparable in terms of the number of treatment modules, intensity, and attention from the treating psychologist.

ELIGIBILITY:
Inclusion Criteria:

* ACS ≥ 6 months before assessment (type 1 MI STEMI/NSTEMI or unstable angina [UA])
* Age 18 and older
* Clinically significant cardiac anxiety that leads to distress and/or interferes with daily life (Cardiac Anxiety Questionnaire; CAQ: ≥18
* Able to read and write in Swedish

Exclusion Criteria:

* Heart failure New York heart Association class IV or ejection fraction ≤ 30%
* Significant valvular disease
* Planned coronary artery bypass surgery or percutaneous interventions
* Any medical restriction to physical exercise
* Severe medical illness or an acute health threatening disease (e.g., cancer)
* Grade 3 hypertension (i.e., blood pressure ≥ 180 systolic and/or 110 diastolic)
* Severe mental illness requiring urgent psychiatric hospitalization or intervention, or risk of suicide
* Alcohol or substance use disorder that would impede ability to complete study protocol
* Ongoing psychological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac anxiety questionnaire modified for weekly assessment | Change over 9 measurement points measured from baseline and weekly for 8 weeks during treatment [PRIMARY ENDPOINT]
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.

SECONDARY OUTCOMES:
Cardiac anxiety questionnaire | From baseline to 8 months
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
Cardiac anxiety questionnaire | From baseline to 1 year and 2 months
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
HeartQoL Health-related Quality of Life Questionnaire modified for weekly assessment | Change over 9 measurement points measured from baseline and weekly for 8 weeks during treatment
  The HeartQoL questionnaire, comprising 14 items, includes a Global scale of 14 items, further divided into Physical (10 items) and Emotional (4 items) subscales. Scores range from 0 to 3, with 3 indicating the highest level and 0 the lowest.
HeartQoL Health-related Quality of Life Questionnaire | From baseline to 8 months
  The HeartQoL questionnaire, comprising 14 items, includes a Global scale of 14 items, further divided into Physical (10 items) and Emotional (4 items) subscales. Scores range from 0 to 3, with 3 indicating the highest level and 0 the lowest.
HeartQoL Health-related Quality of Life Questionnaire | From baseline to 1 year and 2 months
  The HeartQoL questionnaire, comprising 14 items, includes a Global scale of 14 items, further divided into Physical (10 items) and Emotional (4 items) subscales. Scores range from 0 to 3, with 3 indicating the highest level and 0 the lowest.
Symptom checklist Severity and Frequency Scale (SCL, adapted to coronary artery disease) modified for weekly assessment | From baseline to 8 weeks
  Cardiac-related symptoms in two sub scales A) frequency: score ranging from 0-48, with higher score indicating higher frequency of symptoms, B) severity of experienced symptom: score ranging from 0- 48, with a higher score indicating more severe symptoms
Symptom checklist Severity and Frequency Scale (SCL, adapted to coronary artery disease) | From baseline to 8 months
  cardiac-related symptoms in two sub scales A) frequency: score ranging from 0-48, with higher score indicating higher frequency of symptoms, B) severity of experienced symptom: score ranging from 0- 48, with a higher score indicating more severe symptoms
Symptom checklist Severity and Frequency Scale (SCL, adapted to coronary artery disease) | From baseline to 1 year and 2 months
  Cardiac-related symptoms in two sub scales A) frequency: score ranging from 0-48, with higher score indicating higher frequency of symptoms, B) severity of experienced symptom: score ranging from 0- 48, with a higher score indicating more severe symptoms
University of Toronto Atrial fibrillation Severity Scale (AFSS) | Baseline to 8 weeks
  3 item on cardiac-specific healthcare consumption. Scores ranges 0-15 with a higher score indicating more cardiac-related healthcare consumption
University of Toronto Atrial fibrillation Severity Scale (AFSS) | From baseline to 8 months
  3 item on cardiac-specific healthcare consumption. Scores ranges 0-15 with a higher score indicating more cardiac-related healthcare consumption
University of Toronto Atrial fibrillation Severity Scale (AFSS) | From baseline to 1 year and 2 months
  3 item on cardiac-specific healthcare consumption. Scores ranges 0-15 with a higher score indicating more cardiac-related healthcare consumption
Behaviors following cardiac event questionnaire (BCEQ) | From baseline to 8 weeks
  MI-related avoidance questionnaire behaviors developed by the research group
Behaviors following cardiac event questionnaire (BCEQ) | From baseline to 8 months
  MI-related avoidance questionnaire behaviors developed by the research group
Behaviors following cardiac event questionnaire (BCEQ) | From baseline to 1 year and 2 months
  MI-related avoidance questionnaire behaviors developed by the research group
DOSE Non-Adherence questionnaire | From baseline to 8 weeks
  3 items from this two domain scale measuring medical adherence designed to assess missed doses and reasons for missed doses.
DOSE Non-Adherence questionnaire | From baseline to 8 months
  3 items from this two domain scale measuring medical adherence designed to assess missed doses and reasons for missed doses.
DOSE Non-Adherence questionnaire | From baseline to 1 year and 2 months
  3 items from this two domain scale measuring medical adherence designed to assess missed doses and reasons for missed doses.
Perceived stress scale 4-item | Baseline to 8 weeks
  Stress reactivity. A greater score indicate more perceived stress.
Perceived stress scale 4-item | Baseline to 8 months
  Stress reactivity. A greater score indicate more perceived stress.
Perceived stress scale 4-item | Baseline to 1 year and 2 months
  Stress reactivity. A greater score indicate more perceived stress.
Short Fatigue questionnaire | From baseline to 8 weeks
  4-item scale measuring fatigue.
Short Fatigue questionnaire | Baseline to 8 months
  4-item scale measuring fatigue.
Short Fatigue questionnaire | Baseline to 1 year and 2 months
  4-item scale measuring fatigue.
Patient Health Questionnaire-9 | From Baseline to 8 weeks
  Measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression
Patient Health Questionnaire-9 | From Baseline to 8 months
  Measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression
Patient Health Questionnaire-9 | From Baseline to 1 year and 2 months
  Measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression
Insomnia Severity Index | From Baseline to 8 weeks
  Measurement of the degree of sleep difficulties. The total score can range from 0 to 28 points. Higher scores indicate more severe sleep difficulties.
Insomnia Severity Index | From Baseline to 8 months
  Measurement of the degree of sleep difficulties. The total score can range from 0 to 28 points. Higher scores indicate more severe sleep difficulties.
Insomnia Severity Index | From Baseline to 1 year and 2 months
  Measurement of the degree of sleep difficulties. The total score can range from 0 to 28 points. Higher scores indicate more severe sleep difficulties.
Perceived stress scale 4-item | Change over 9 measurement points measured from baseline and weekly for 8 weeks during treatment
  Stress reactivity. A greater score indicate more perceived stress.
The Godin Leisure-time Exercise and International Physical Activity Questionnaire 1 item on inactivity | Baseline to 8 weeks
  Level of physical activity and inactivity: On the Godin leisure-time excercise: The participant rate numbers of time per week that they engage in physical activity. The numb ers are the categorized in to low, moderate, and high levels of physical activity. And from International Physical Activity Questionnaire we will use 1 item on inactivity
The Godin Leisure-time Exercise and International Physical Activity Questionnaire 1 item on inactivity | Baseline to 8 months
  Level of physical activity and inactivity: On the Godin leisure-time excercise: The participant rate numbers of time per week that they engage in physical activity. The numb ers are the categorized in to low, moderate, and high levels of physical activity. And from International Physical Activity Questionnaire we will use 1 item on inactivity
The Godin Leisure-time Exercise and International Physical Activity Questionnaire 1 item on inactivity | Baseline to 1 year and 2 months
  Level of physical activity and inactivity: On the Godin leisure-time excercise: The participant rate numbers of time per week that they engage in physical activity. The numb ers are the categorized in to low, moderate, and high levels of physical activity. And from International Physical Activity Questionnaire we will use 1 item on inactivity
Lifestyle factors: The national Board of health and Welfare questionnaire | Baseline to 8 weeks
  Questionnaire regarding diet (5 item), tobacco (2 item) and alcohol (3 item) diet (5 item), tobacco (2 item) and alcohol (3 item) and BMI.
Lifestyle factors: The national Board of health and Welfare questionnaire | Baseline to 8 months
  Questionnaire regarding diet (5 item), tobacco (2 item) and alcohol (3 item) diet (5 item), tobacco (2 item) and alcohol (3 item) and BMI.
Lifestyle factors: The national Board of health and Welfare questionnaire | Baseline to 1 year and 2 months
  Questionnaire regarding diet (5 item), tobacco (2 item) and alcohol (3 item) diet (5 item), tobacco (2 item) and alcohol (3 item) and BMI.
Aversive cognition to medication | Baseline to 8 weeks
  : A 3-item subset of questions with regards to psychological distress associated with cardiac medication
Adversive cognition to medication | Baseline to 8 months
  : A 3-item subset of questions with regards to psychological distress associated with cardiac medication
Adversive cognition to medication | Baseline to 1 year and 2 months
  : A 3-item subset of questions with regards to psychological distress associated with cardiac medication

OTHER OUTCOMES:
Adverse events | Baseline to 8 weeks
  Potential adverse reactions to the treatment. Participants will be asked to report and rate
Adverse events | Baseline to 8 months
  Potential adverse reactions to the treatment. Participants will be asked to report and rate
Adverse events | Baseline to 1 year and 2 months
  Potential adverse reactions to the treatment. Participants will be asked to report and rate
Adverse events | Change over 9 measurement points measured from baseline and weekly for 8 weeks during treatment
  Potential adverse reactions to the treatment. Participants will be asked to report and rate
Accelerometer (Actigraf®) | Baseline to 8 weeks
  n Accelerometer (Actigraf®) will be carried on the wrist over to measure physical activity over 1 week
Accelerometer (Actigraf®) | Baseline to 1 year and 2 months
  n Accelerometer (Actigraf®) will be carried on the wrist over to measure physical activity over 1 week
Swedish Prescribed Drug Register | Retrospective period of 6 months at baseline
  The prescription fill-rate of cardiovascular medication (e.g., statin)will be collected and will be used to calculate the proportion of days covered (PDC) with a statin. A PDC <80% will be used to indicate nonadherence as per convention in other studies of cardiovascular medication refills.
Swedish Prescribed Drug Register | Retrospective period from 6 months at 6 month follow up
  The prescription fill-rate of cardiovascular medication (e.g., statin)will be collected and will be used to calculate the proportion of days covered (PDC) with a statin. A PDC <80% will be
Swedish Prescribed Drug Register | Retrospective period from 6 months at 12 month follow up
  The prescription fill-rate of cardiovascular medication (e.g., statin)will be collected and will be used to calculate the proportion of days covered (PDC) with a statin. A PDC <80% will be
Working Alliance Inventory | 2 weeks from baseline
  Measures therapeutic alliance with the psychologist
Treatment Credibility Scale | Measures treatment credibility
  2 weeks from baseline
Client satisfaction Questionnaire | Baseline to 8 weeks
  Treatment satisfaction, score ranging from 0 to 32, with a higher score indication more satisfaction with the treatment.
Follow-up questions on health changes | Baseline to 8 weeks
  We will ask participant to describe if they have experienced any psychosocial stressors, changes in physical health, such as invasive therapy and changes of medication
Follow-up questions on health changes | Baseline to 8 months
  We will ask participant to describe if they have experienced any psychosocial stressors, changes in physical health, such as invasive therapy and changes of medication
Follow-up questions on health changes | Baseline to 1 year and 2 months
  We will ask participant to describe if they have experienced any psychosocial stressors, changes in physical health, such as invasive therapy and changes of medication
AFFS/SCL-4 | Change over 9 measurement points measured from baseline and weekly for 8 weeks during treatment
  4 items derived from the Symptoms Checklist (SCL) and the Atrial Fibrillation Severity Scale (AFSS) measuring disabling cardiac symptoms
Behaviors following cardiac event questionnaire (BCEQ) | Change over 9 measurement points measured from baseline and weekly for 8 weeks during treatment
  5 items measuring avoidance behavior from the MI-related avoidance questionnaire behaviors developed by the research group
DOSE Non-Adherence questionnaire | Change over 9 measurement points measured from baseline and weekly for 8 weeks during treatment
  3 items from this two domain scale measuring medical adherence designed to assess missed doses and reasons for missed doses.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
The individual participant data underlying the analyses in this study cannot be made publicly available due to Swedish and European Union data protection regulations. Requests for additional outcomes or estimates may be directed to the corresponding author and will be handled in accordance with legal expertise and the sponsor's current data governance guidelines

REFERENCES:
- [Derived] Johnsson A, Ljotsson B, Braunschweig F, Mellbin LG, Sarnholm J. Digital cognitive behavioural therapy for cardiac anxiety following acute coronary syndrome: protocol for a randomised controlled trial comparing CBT to a digital lifestyle intervention. BMJ Open. 2025 Oct 28;15(10):e106473. doi: 10.1136/bmjopen-2025-106473. PMID 41151962